CLINICAL TRIAL: NCT05813223
Title: The Effect of Acute and Prolonged Administration of Gefapixant on Cough-related Brain Activity in Patients With Chronic Cough
Brief Title: Effect of Gefapixant on Cough-related Brain Activity in Patients With Chronic Cough
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stuart Mazzone (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Melbourne Health (Other); Monash University (Other)
Responsible Party: Sponsor-Investigator, Stuart Mazzone, Professor, University of Melbourne
Organization: University of Melbourne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023.005
Record Dates: First submitted 2023-03-20; First posted 2023-04-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Cough
Keywords: functional brain imaging; ATP; Capsaicin; Refractory chronic cough; Mechanism of Disease
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Intervention Model Description: Open label, single arm, mechanism of disease study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gefapixant treatment (Experimental): Participants will asked to take an oral tablet containing 45mg Gefapixant twice daily (BID).
  Interventions: Drug: Gefapixant

INTERVENTIONS:
Drug: Gefapixant — Purinergic (P2X3) Receptor antagonist. Film-coated tablet taken orally.
  Other Names: Merck (MK)-7264

SUMMARY:
Recently, a new drug called Gefapixant passed phase III clinical trials for cough suppression in patients with chronic cough. The goal of this clinical trial is to investigate the effect of acute and prolonged administration of the drug Gefapixant on cough-related brain activity in patients with chronic cough. The main question it aims to answer is: does the mechanism of action of Gefapixant on the brainstem and brain circuits regulating cough differ between acute and prolonged therapy in people with chronic cough?

Participants have their brain activity and their sensitivity to cough-inducing substances measured as well as complete questionnaires about their cough before and while taking daily Gefapixant.

DETAILED DESCRIPTION:
Chronic cough is a distressing disorder experienced by 1 in 10 people worldwide. At its worst, individuals can cough hundreds of times every hour of their waking lives, and this can persist for decades without relief. Chronic cough sufferers also experience an ongoing feeling of needing to cough (urge-to-cough) that prompts coughing and throat clearing, but usually without resolution of the sensation. The clinical problem is extremely challenging to manage because the last dedicated cough suppressant drug to be approved for clinical use (dextromethorphan) was in 1958 and it offers no benefit for chronic cough patients.

Recently, a new drug called Gefapixant passed phase III clinical trials for cough suppression in patients with chronic cough and is currently advancing to market globally. Gefapixant is extremely well-tolerated with minimal side effects - a reduction in taste acuity being the main adverse effect reported. This project will investigate further the mechanisms of action of Gefapixant, assessing for the first time the effects of Gefapixant therapy on the brain pathways involved in cough and urge-to-cough generation.

The study will recruit 31 participants with existing chronic cough and investigate their brain responses using non-invasive magnetic resonance imaging while briefly breathing personally tailored stimuli that are just below threshold for triggering coughing (determined using inhaled cough challenge testing procedures). Brain scans will be performed before and at two time points (3 days and 12 weeks) after starting Gefapixant treatment, consisting of one 45mg tablet swallowed twice daily.

Participants will also complete questionnaires and maintain a diary about their cough. After 12 weeks of treatment, participants will cease taking Gefapixant for 1 week and brain scans will be performed again to assess whether changes in brain activity are sustained. Participants will then have access to Gefapixant for a further 9 months during which time cough sensitivity and questionnaires and will be assessed on 2 additional occasions to determine whether longer term therapy leads to added changes in nerve pathways mediating cough.

Significance: Understanding how the brain controls cough and the urge-to-cough, and the specific brain processes altered by Gefapixant therapy, will significantly advance the understanding of the biology and clinical management of this challenging clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study. 18-65 years old; Male or female.
* Non-smokers for at least 5 years and have no history of neurological disease or any recent history (over 8 weeks) of acute respiratory infections.
* Presence of Refractory Chronic Cough (RCC) or Unexplained Chronic Cough (UCC) for ≥1 year, defined as cough unresponsive to treatment for underlying conditions including reflux disease, asthma and rhinitis.
* Presence of cough symptoms as determined by a self-reported cough severity of ≥40mm on 10-point scale on screening.

Exclusion Criteria:

* Current smokers or recreational drug users.
* Women who are pregnant.
* People with contraindications to MRI scanning (i.e. metal implants, claustrophobia).
* Children and/or young people (ie. <18 years).
* People with an intellectual or mental impairment.
* People highly dependent on medical care.
* People in existing dependent or unequal relationships with any member of the research team.
* People with known allergy to chili (very rare).
* Non-English speakers (as English proficiency is required to accurately complete research tasks).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cough-related brain activity using brain imaging following Gefapixant administration | Gefapixant administration will be for 12 weeks with brain scans to be performed before, 3 days after, and 12 weeks after dosing.
  We will investigate the time-dependent effect of Gefapixant treatment on brain activity evoked by inhaled ATP and capsaicin as measured using functional Magnetic Resonance Imaging (fMRI). The principle endpoint is measured as the change in capsaicin and ATP evoked Blood Oxygen Level Dependent (BOLD) signal and the unit of measure is percentage.
Change in cough-related brain activity using brain imaging following Gefapixant withdrawal | Brain imaging will be performed 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing and investigate the time-dependent effect of Gefapixant treatment on brain activity evoked by inhaled ATP and capsaicin as measured using functional Magnetic Resonance Imaging (fMRI). The principle endpoint is measured as the change in capsaicin and ATP evoked Blood Oxygen Level Dependent (BOLD) signal and the unit of measure is percentage.

SECONDARY OUTCOMES:
Change in capsaicin and ATP cough challenge test sensitivity following Gefapixant administration | Cough thresholds will be determined before, 3 days after and 12 weeks after Gefapixant dosing.
  We will investigate participant's cough sensitivity thresholds by inhaled cough challenge testing. This involves participants inhaling single breaths of increasing concentrations of tussigenic stimuli (capsaicin and ATP) as well as saline control to determine threshold doses that elicit an urge to cough, two coughs (C2) and five coughs (C5). The principle endpoint is measured as the change in capsaicin and ATP concentration needed to elicit cough responses and the unit of measure is micromolar.
Change in Urge To Cough Visual Analogue Scale (UTCVAS) score after Gefapixant administration | Participant self-reports using the UTCVAS will be collected before and 3 days, 4 weeks, 8 weeks and 12 weeks after Gefapixant dosing.
  Participants will be asked to self-report on their urge to cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No urge to cough" and a maximum value of 100 labelled "Worst urge to cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in UTCVAS score and the unit of measure is points.
Change in Cough Visual Analogue Scale (CVAS) score after Gefapixant administration | Participant self-reports using the CVAS will be collected before and 3 days, 4 weeks, 8 weeks and 12 weeks after Gefapixant dosing.
  Participants will be asked to self-report on their cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No cough" and a maximum value of 100 labelled "Worst cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in CVAS score and the unit of measure is points.
Change in Leicester Cough Questionnaire (LCQ) score after Gefapixant administration | Participant self-reports using the LCQ will be collected before and 3 days, 4 weeks, 8 weeks and 12 weeks after Gefapixant dosing.
  Participants will be asked to self-report on the impact of cough on their quality of life. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to the impact of cough in one of three domains (physical, psychological social). The LCQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in LCQ score and the unit of measure is points.
Change in Newcastle Laryngeal Hypersensitivity Questionnaire (NLHQ) score after Gefapixant administration | Participant self-reports using the NLHQ will be collected before and 3 days, 4 weeks, 8 weeks and 12 weeks after Gefapixant dosing.
  Participants will be asked to self-report on sensations related to laryngeal hypersensitivity. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to an upper airway sensation in one of three domains (throat obstruction, throat pain/thermal), throat tickle). The NHLQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in NLHQ score and the unit of measure is points.
Change in Hull Airway Reflux Questionnaire (HARQ) score after Gefapixant administration | Participant self-reports using the HARQ will be collected before and 3 days, 4 weeks, 8 weeks and 12 weeks after Gefapixant dosing.
  Participants will be asked to self-report on symptoms related to airway reflux. Each item requires a rating on a 6-point Likert scale from 0 to 5 and is related to an aspect of airway reflux. The HARQ is scored by adding the total ratings (range 0-70). A higher score indicates a worse outcome. The principal endpoint is measured as the change in HARQ score and the unit of measure is points.
Change in Cough Severity Diary (CSD) score after Gefapixant administration | Participant self-reports using the CSD will be collected every day for 12 weeks after the start of Gefapixant administration.
  Participants will be asked to self-report on their daily cough severity. Each item requires a rating on an 11-point Likert scale from 0 to 10 and is related to an aspect of cough in one of three domains (frequency, intensity, disruption). The CSD is scored by averaging the ratings in each domain, as well as averaging across all items (range 1-10). A higher score indicates a worse outcome. The principal endpoint is measured as the change in CSD score and the unit of measure is points.
Change in capsaicin and ATP cough challenge test sensitivity following Gefapixant withdrawal | Cough thresholds will be determined 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing and investigate participant's cough sensitivity thresholds by inhaled cough challenge testing. This involves participants inhaling single breaths of increasing concentrations of tussigenic stimuli (capsaicin and ATP) as well as saline control to determine threshold doses that elicit an urge to cough, two coughs (C2) and five coughs (C5). The principle endpoint is measured as the change in capsaicin and ATP concentration needed to elicit cough responses and the unit of measure is micromolar.
Change in Urge To Cough Visual Analogue Scale (UTCVAS) score following Gefapixant withdrawal | Participant self-report using the UTCVAS will be collected 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on their urge to cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No urge to cough" and a maximum value of 100 labelled "Worst urge to cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in UTCVAS score and the unit of measure is points.
Change in Cough Visual Analogue Scale (CVAS) score following Gefapixant withdrawal | Participant self-report using the CVAS will be collected 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on their cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No cough" and a maximum value of 100 labelled "Worst cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in CVAS score and the unit of measure is points.
Change in Leicester Cough Questionnaire (LCQ) score following Gefapixant withdrawal | Participant self-report using the LCQ will be collected 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on the impact of cough on their quality of life. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to the impact of cough in one of three domains (physical, psychological social). The LCQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in LCQ score and the unit of measure is points.
Change in Newcastle Laryngeal Hypersensitivity Questionnaire (NLHQ) score following Gefapixant withdrawal | Participant self-report using the NHLQ will be collected 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on sensations related to laryngeal hypersensitivity. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to an upper airway sensation in one of three domains (throat obstruction, throat pain/thermal), throat tickle). The NHLQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in NLHQ score and the unit of measure is points.
Change in Hull Airway Reflux Questionnaire (HARQ) score following Gefapixant withdrawal | Participant self-report using the HARQ will be collected 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on symptoms related to airway reflux. Each item requires a rating on a 6-point Likert scale from 0 to 5 and is related to an aspect of airway reflux. The HARQ is scored by adding the total ratings (range 0-70). A higher score indicates a worse outcome. The principal endpoint is measured as the change in HARQ score and the unit of measure is points.
Change in Cough Severity Diary (CSD) score following Gefapixant withdrawal | Participant self-report using the CSD will be collected every day in the 1 week after Gefapixant withdrawal (Week 13).
  We will follow up with participants 1 week after stopping Gefapixant dosing. Participants will be asked to self-report on their daily cough severity. Each item requires a rating on an 11-point Likert scale from 0 to 10 and is related to an aspect of cough in one of three domains (frequency, intensity, disruption). The CSD is scored by averaging the ratings in each domain, as well as averaging across all items (range 1-10). A higher score indicates a worse outcome. The principal endpoint is measured as the change in CSD score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on cough challenge sensitivity. | Cough thresholds will be determined at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. We will investigate participant's cough sensitivity thresholds by inhaled cough challenge testing. This involves participants inhaling single breaths of increasing concentrations of tussigenic stimuli (capsaicin and ATP) as well as saline control to determine threshold doses that elicit an urge to cough, two coughs (C2) and five coughs (C5). The principle endpoint is measured as the change in capsaicin and ATP concentration needed to elicit cough responses and the unit of measure is micromolar.
Sustainability of Gefapixant treatment effects on Urge To Cough Visual Analogue Scale (UTCVAS) score | Participant self-report using the UTCVAS will be collected at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on their urge to cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No urge to cough" and a maximum value of 100 labelled "Worst urge to cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in UTCVAS score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on Cough Visual Analogue Scale (CVAS) score | Participant self-report using the CVAS will be collected at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on their cough severity using the Urge to Cough Visual Analogue Scale. The scale is 100 units with a minimum value of 0 labelled "No cough" and a maximum value of 100 labelled "Worst cough ever". A higher score indicates a worse outcome. The principal endpoint is measured as the change in CVAS score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on Leicester Cough Questionnaire (LCQ) score | Participant self-report using the LCQ will be collected at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on the impact of cough on their quality of life. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to the impact of cough in one of three domains (physical, psychological social). The LCQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in LCQ score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on Newcastle Laryngeal Hypersensitivity Questionnaire (NLHQ) score | Participant self-report using the NLHQ will be collected at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on sensations related to laryngeal hypersensitivity. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to an upper airway sensation in one of three domains (throat obstruction, throat pain/thermal), throat tickle). The NHLQ is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the change in NLHQ score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on Hull Airway Reflux Questionnaire (HARQ) score | Participant self-report using the HARQ will be collected at 6 and 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on symptoms related to airway reflux. Each item requires a rating on a 6-point Likert scale from 0 to 5 and is related to an aspect of airway reflux. The HARQ is scored by adding the total ratings (range 0-70). A higher score indicates a worse outcome. The principal endpoint is measured as the change in HARQ score and the unit of measure is points.
Sustainability of Gefapixant treatment effects on Cough Severity Diary (CSD) score | Participant self-report using the CSD will be collected every day from Week 14 until 12 months (relative to start of study).
  Participants can opt to resume Gefapixant administration for another 9 months after completion of the withdrawal assessments. Participants will be asked to self-report on their daily cough severity. Each item requires a rating on an 11-point Likert scale from 0 to 10 and is related to an aspect of cough in one of three domains (frequency, intensity, disruption). The CSD is scored by averaging the ratings in each domain, as well as averaging across all items (range 1-10). A higher score indicates a worse outcome. The principal endpoint is measured as the change in CSD score and the unit of measure is points.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart B Mazzone, PhD, Principal Investigator — +61383446457
Locations (1):
- The University of Melbourne, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung KF, Pavord ID. Prevalence, pathogenesis, and causes of chronic cough. Lancet. 2008 Apr 19;371(9621):1364-74. doi: 10.1016/S0140-6736(08)60595-4. PMID 18424325
- [Background] Chung KF, McGarvey L, Mazzone SB. Chronic cough as a neuropathic disorder. Lancet Respir Med. 2013 Jul;1(5):414-22. doi: 10.1016/S2213-2600(13)70043-2. Epub 2013 May 3. PMID 24429206
- [Background] Mazzone SB, McLennan L, McGovern AE, Egan GF, Farrell MJ. Representation of capsaicin-evoked urge-to-cough in the human brain using functional magnetic resonance imaging. Am J Respir Crit Care Med. 2007 Aug 15;176(4):327-32. doi: 10.1164/rccm.200612-1856OC. Epub 2007 Jun 15. PMID 17575093
- [Background] Ando A, Smallwood D, McMahon M, Irving L, Mazzone SB, Farrell MJ. Neural correlates of cough hypersensitivity in humans: evidence for central sensitisation and dysfunctional inhibitory control. Thorax. 2016 Apr;71(4):323-9. doi: 10.1136/thoraxjnl-2015-207425. Epub 2016 Feb 9. PMID 26860344
- [Background] Thomas D, Gibson PG. Gefapixant for chronic cough. Lancet. 2022 Mar 5;399(10328):886-887. doi: 10.1016/S0140-6736(21)02438-7. No abstract available. PMID 35248173
- [Background] McGarvey LP, Birring SS, Morice AH, Dicpinigaitis PV, Pavord ID, Schelfhout J, Nguyen AM, Li Q, Tzontcheva A, Iskold B, Green SA, Rosa C, Muccino DR, Smith JA; COUGH-1 and COUGH-2 Investigators. Efficacy and safety of gefapixant, a P2X3 receptor antagonist, in refractory chronic cough and unexplained chronic cough (COUGH-1 and COUGH-2): results from two double-blind, randomised, parallel-group, placebo-controlled, phase 3 trials. Lancet. 2022 Mar 5;399(10328):909-923. doi: 10.1016/S0140-6736(21)02348-5. PMID 35248186
- [Background] Smith JA, Kitt MM, Morice AH, Birring SS, McGarvey LP, Sher MR, Li YP, Wu WC, Xu ZJ, Muccino DR, Ford AP; Protocol 012 Investigators. Gefapixant, a P2X3 receptor antagonist, for the treatment of refractory or unexplained chronic cough: a randomised, double-blind, controlled, parallel-group, phase 2b trial. Lancet Respir Med. 2020 Aug;8(8):775-785. doi: 10.1016/S2213-2600(19)30471-0. Epub 2020 Feb 25. PMID 32109425
- [Background] Morice AH, Jakes AD, Faruqi S, Birring SS, McGarvey L, Canning B, Smith JA, Parker SM, Chung KF, Lai K, Pavord ID, van den Berg J, Song WJ, Millqvist E, Farrell MJ, Mazzone SB, Dicpinigaitis P; Chronic Cough Registry. A worldwide survey of chronic cough: a manifestation of enhanced somatosensory response. Eur Respir J. 2014 Nov;44(5):1149-55. doi: 10.1183/09031936.00217813. Epub 2014 Sep 3. PMID 25186267
- [Background] Morice AH, Kitt MM, Ford AP, Tershakovec AM, Wu WC, Brindle K, Thompson R, Thackray-Nocera S, Wright C. The effect of gefapixant, a P2X3 antagonist, on cough reflex sensitivity: a randomised placebo-controlled study. Eur Respir J. 2019 Jul 4;54(1):1900439. doi: 10.1183/13993003.00439-2019. Print 2019 Jul. PMID 31023843
- [Background] Dicpinigaitis PV, Alva RV. Safety of capsaicin cough challenge testing. Chest. 2005 Jul;128(1):196-202. doi: 10.1378/chest.128.1.196. PMID 16002935